CLINICAL TRIAL: NCT02864277
Title: Enhanced Recovery After Surgery (ERAS) Program Versus Conventional Perioperative Strategies in Patients Undergoing Gynecologic Oncologic Surgery: A Randomized Controlled Trial
Brief Title: Enhanced Recovery After Surgery Gynecology Oncology
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00203177
Record Dates: First submitted 2016-07-11; First posted 2016-08-12 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Malignant Female Reproductive System Neoplasm
Keywords: Gynecology; Cancer; General Surgery; Recovery Quality; Length of hospital stay
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention Conventional Strategy (No Intervention): Perioperative Anesthetic No Intervention Management: Conventional Strategy Group 4 pages of concise directions on how to take care of the participant.
- ERAS Group (Experimental): ERAS (enhanced recovery after surgery)
  Interventions: Procedure: No Intervention Conventional Strategy; Procedure: ERAS

INTERVENTIONS:
Procedure: No Intervention Conventional Strategy — The Conventional Strategy Group description encompasses over 4 pages of concise directions on how to take care of the participant. This cannot be reduced to less than 1000 characters.
  Preoperative Management Interoperative Management Postoperative Management Post discharge
  Arms: ERAS Group
Procedure: ERAS — The ERAS Group description encompasses over 3 pages of concise directions on how to take care of the participant. This cannot be reduced to less than 1000 characters.
  Preoperative Management Interoperative Management Postoperative Management Post discharge
  Arms: ERAS Group

SUMMARY:
The aim of this study is to compare outcomes of conventional perioperative care with those of an enhanced recovery after surgery (ERAS) perioperative care plan in women undergoing open abdominal surgery for gynecologic cancer or suspected gynecologic cancer. Investigators hypothesize that those patients randomized to the ERAS protocol will have shorter lengths of hospital stay, without increasing readmission rates. ASD

DETAILED DESCRIPTION:
The study design is a two-arm, randomized, controlled trial. The control arm will consist of standard conventional perioperative care. The intervention arm will consist of a protocol-driven ERAS program. All patients with a known or suspected gynecologic malignancy scheduled for open abdominal surgery from the gynecologic oncology clinic will be screened for study eligibility. Those eligible for the study will be approached for participation in the study and provided written informed consent.

Once enrolled, study participants will be randomized into two arms (control group and ERAS group) using block randomization (block size=6). Block randomization will be performed using an online randomization generator that can be accessed at http://www.sealed envelope.com/simple randomizer /v1/lists . Due to the requirement for active patient and provider participation, it will not be possible to perform the study with blinded participants and care providers. Study investigators responsible for data collection and outcomes assessment will be blinded to randomization assignments. Once randomized, patients will be seen in preoperative clinic and given specific preoperative instructions as dictated by their study group.

On the day of surgery, patients will receive perioperative care as per protocol, based on their assigned group.

During postoperative care, patients will be asked to fill out a daily diary to document their recovery progress, where they will assess their ability to meet the study milestones, as noted above (e.g. pain and ambulation).

Patients will be eligible for discharge once meeting all pre-defined discharge criteria, including: tolerating oral fluid and diet, pain controlled with oral pain regimen, have return of bowel function (flatus), are self-caring (able to dress, shower, and groom themselves), and are mobilizing independently. Assessment of these parameters will be made by gynecologic oncology clinicians.

After discharge, patients will follow-up in gynecologic oncology clinic at 2 weeks and 6 weeks postoperatively.

Both arms of the study will be protocol-driven, with checklists for patients, nursing staff, and house staff to help with compliance. Teaching sessions and dry runs will be held before trial commencement to clarify points of confusion and to reduce protocol violations.

Data collection on subjects will be performed throughout the duration of their enrollment in the study. Data will be abstracted for medical record charts from Enterprise Data Warehouse and corroborated with Power chart (Northwestern Memorial Hospital), EPIC (Northwestern Memorial Hospital Medical record system), and Surginet (Northwestern Memorial Hospital Surgical Medical Record System).

In addition to the demographic and clinical information that will be abstracted from the medical record, subjects will also complete a validated Quality of Recovery Survey (the QOR (Quality of Recovery-40 question survey) at 2 weeks post-surgery. Lastly, C-Reactive Protein (CRP) and Interleukin-6 (IL-6) levels will be determined from blood collected pre-operatively (to coincide with scheduled pre-operative clinic visit) and on post-operative day 1 (POD#1 (post operative day )], to coincide with scheduled POD#1 blood draw). Blood samples will be collected in provided, 10ml red topped vacuum collection tubes (no anti-coagulant). After collection of the whole blood, the blood will be allowed to clot by leaving it undisturbed at room temperature for 30 minutes. Clot will be removed by centrifugation at 2,000 x g for 10 minutes in a 4°C refrigerated centrifuge. Using a Pasteur pipette the liquid supernatant (serum) will be immediately transferred to collection tube and apportioned into 0.5 ml aliquots and frozen in liquid nitrogen. Samples will be batch processed for CRP and IL-6 levels by ELISA according to manufacturer instructions (affymetrix eBioscience Catalog Numbers: 88-7502 and 88-7066).

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-70 years
* Fluent in English language
* Known or suspected diagnosis of gynecologic malignancy (including ovarian, endometrial, and cervical cancers)
* Scheduled for elective laparotomy
* Medically eligible for major surgical procedure

Exclusion Criteria:

* Unable to mobilize independently preoperatively
* The following populations will not be included in the study: adults unable to consent (such as the cognitively impaired), minors < 18 years of age, pregnant women, and prisoners.
* Emergency surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Total length of hospital stay (days) | Up to 10 days
  total length of hospital stay (days)

SECONDARY OUTCOMES:
Achievement of Postoperative Milestones | 30 days
  Achievement of the below milestones:
  A) Void Freely(Return of Bladder Function) B) Pain Controlled with oral Medications C) Eating Target Diet without emesis D) Passing Flatus (Return of Bowel Function) E) Ambulating at Baseline F) Self Care at Baseline
Surgical complications | 30 days
  Surgical complications within 30 days of procedure
Readmission rates | 2 week and 30 day
  Readmission rates assessed at 2 week and 30 day
Time to adjuvant treatment | 60 days
  Time participant receives adjuvant treatment, if needed (chemotherapy or radiation)
30-day mortality rates | 30 days
  30-day mortality rates of participants
Patient reported satisfaction | 14 days
  Quality of Recovery 40 questionnaire results from participants
Progression-free survival | 2 years
  Progression-free survival post procedure
Preoperative vs postoperative day # 1 C-Reactive Protein (CRP) | 24 hours post surgery
  Preoperative vs postoperative day #1 C-Reactive Protein (CRP) levels for all participants blood samples.
Preoperative vs postoperative day # 1 Interleukin-6 (IL-6) levels | 24 hours post surgery
  Preoperative vs postoperative day #1 Interleukin-6 (IL-6) levels for all participants blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Shireen Ahmad, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tewari KS, Java JJ, Eskander RN, Monk BJ, Burger RA. Early initiation of chemotherapy following complete resection of advanced ovarian cancer associated with improved survival: NRG Oncology/Gynecologic Oncology Group study. Ann Oncol. 2016 Jan;27(1):114-21. doi: 10.1093/annonc/mdv500. Epub 2015 Oct 20. PMID 26487588
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Lu D, Wang X, Shi G. Perioperative enhanced recovery programmes for gynaecological cancer patients. Cochrane Database Syst Rev. 2015 Mar 19;2015(3):CD008239. doi: 10.1002/14651858.CD008239.pub4. PMID 25789452
- [Background] Nelson G, Kalogera E, Dowdy SC. Enhanced recovery pathways in gynecologic oncology. Gynecol Oncol. 2014 Dec;135(3):586-94. doi: 10.1016/j.ygyno.2014.10.006. Epub 2014 Oct 12. PMID 25316179
- [Background] Wijk L, Franzen K, Ljungqvist O, Nilsson K. Implementing a structured Enhanced Recovery After Surgery (ERAS) protocol reduces length of stay after abdominal hysterectomy. Acta Obstet Gynecol Scand. 2014 Aug;93(8):749-56. doi: 10.1111/aogs.12423. Epub 2014 Jun 13. PMID 24828471
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396